CLINICAL TRIAL: NCT02160301
Title: Effect of a Multimodal Pain Regimen on Pain Control, Patient Satisfaction and Narcotic Use in Orthopaedic Trauma Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient infrastructure/funding for enrollment
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2669
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Post Operative Pain Control
Keywords: pain; postoperative; multimodal; satisfaction; narcotic
MeSH Terms: conditions — Pain; Personal Satisfaction | interventions — Gabapentin; Acetaminophen; Celecoxib; Dexamethasone; Calcium Dobesilate; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multimodal pain control (Experimental): Oxycodone 5-15mg PO q4hrs prn pre- and post-op, Acetaminophen 1000mg IV once pre-op, Acetaminophen 1000mg PO q8hrs pre-op and x2 weeks post op, prn thereafter, Gabapentin 100mg/200mg PO a8hrs pre-op and x2 weeks post op, Dexamethasone 8mg IV once intra-op, Celecoxib 400mg PO once pre-op.
  Interventions: Drug: Gabapentin; Drug: Acetaminophen; Drug: Celecoxib; Drug: Dexamethasone; Drug: Oxycodone
- Standard pain control (Active Comparator): Oxycodone 5-15mg PO q4hrs prn, Acetaminophen 1000mg PO q8hrs prn.
  Interventions: Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Gabapentin — PO
  Other Names: Neurontin
  Arms: Multimodal pain control
Drug: Acetaminophen — PO
  Other Names: Tylenol; Acephen; Cetafen; Mapap; Q-Pap; Valorin
Drug: Acetaminophen — IV
  Other Names: Ofirmev
  Arms: Multimodal pain control
Drug: Celecoxib — PO
  Other Names: Celebrex
  Arms: Multimodal pain control
Drug: Dexamethasone — IV
  Other Names: Baycadron
  Arms: Multimodal pain control
Drug: Oxycodone — PO
  Other Names: Roxicodone

SUMMARY:
The study is a prospective, randomized, open-label comparison of a multimodal regimen and a standard, narcotic-based regimen for postoperative pain control in patients undergoing surgery for an operatively indicated, isolated extremity fracture. The investigators will be measuring pain levels, narcotic use, patient satisfaction, patient reported function, adverse events and fracture union. The investigators hypothesize that this multimodal regimen will lead to improved pain, less narcotic use and improved satisfaction as compared to the standard regimen.

DETAILED DESCRIPTION:
Patients will be assessed for inclusion or exclusion during admission to the hospital or during evaluation in the clinic or emergency room for an isolated extremity fracture for which surgery is indicated. Once enrolled in the study and consent obtained, patients will be randomized into either the standard therapy group or the multimodal therapy group using permuted block randomization based on injury site. The sites of fracture are as follows:

* wrist/hand/forearm
* elbow/upper arm/shoulder
* acetabulum/pelvis
* foot/ankle
* patella/tibia (shaft, proximal)
* femur (proximal to distal)

The investigators have assumed that these distinct areas result in a similar amount of disability and pain as compared to the other sites. This is an attempt to mitigate the possible confounder of disproportionate numbers of more painful or more debilitating injuries falling in one study group compared to another.

Pre-operatively, patient demographic data will be recording including age, gender, BMI, hand dominance, occupation, use of tobacco/alcohol/illicit drugs, use of assistive devices, relevant comorbidities (i.e., diabetes), site of injury, mechanism and energy (high or low). If there is to be a delay between initial presentation and surgery, as is often the case for distal radius or ankle fractures, among others, multimodal patients will begin their therapy immediately after evaluation. Thus, they will be started on scheduled 1000mg acetaminophen and 100mg gabapentin both three times daily. They will also be provided an 5mg oxycodone prescription with instructions to take 1-3 tablets every 4 hours as needed for pain. Standard therapy patients will be prescribed oxycodone alone, using the same parameters, with the ability to take acetaminophen on an as needed basis.

Pre-operatively, multimodal patients will receive 1000mg IV acetaminophen, 100mg PO gabapentin and 400mg PO celecoxib. All patients will have a peripheral nerve block placed when indicated, to confirm to the investigators standard of care. Patients will then undergo surgery with the investigators standardized anesthesia protocol as described in the protocol. Intraoperatively, multimodal patients will receive 8mg of IV dexamethasone. Post-operatively, multimodal patients will be given 1000mg acetaminophen three times daily for the duration of their narcotic use and 100mg Gabapentin three times daily for 1 week, which will be titrated to 200mg three times daily for 1 additional week. They will also receive an oxycodone prescription as described previously. Standard therapy patients will be given an oxycodone prescription alone with the advice to take tylenol on an as needed basis not to exceed 4000mg/day. No placebo medications will be used as this is an open label study.

Patients will be instructed to avoid all anti-inflammatory medications. All patients across groups will be given aspirin 81mg for deep vein thrombosis prophylaxis if they suffered a lower extremity fracture. Should a patient require an alternative deep vein thrombosis prophylaxis regimen due to an allergy to aspirin or a personal history of deep vein thromboses, low molecular weight heparin will be used.

Patients will be given a diary to record their daily narcotic use, daily minimum, maximum and average pain scores using a visual analog scale and any side effects. Patients will be provided the contact information of the attending surgeon's nurse to report any serious allergies or adverse effects of the study medications. A case by case decision will be made to either continue the protocol or to drop the patient from the study and make needed medications changes.

Patients will be followed at defined time points after surgery including, 2 wks, 6wks, 3mo and 6mo.

At their 2 wk follow up visit they will fill out the Short Musculoskeletal Function Assessment for their preoperative functional state as well as the American Pain Society Patient Satisfaction Questionnaire. These will again be filled out at their 3 and 6 month visits. Union will be assessed at their 3 and 6 month visits by a third party, blinded observed. It will be defined as three cortices of bridging callus on 2 orthogonal views. Once fracture union occurs or nonunion is identified control patients will be allowed to use non steroidal anti-inflammatories as needed. Time to return to work/normal activity, total narcotic usage and duration of narcotic use will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Bone fracture
* Isolated injury
* Requires operative intervention

Exclusion Criteria:

* pathological fractures
* inability to personally consent to participation due to cognitive impairment, intoxication or sedation
* severe head injury
* polytrauma patients with multiple fractures or other injuries
* pregnancy
* open fractures
* metabolic bone disease
* allergies or contraindications to the study medications, including sulfa medications.
* prior or current drug or alcohol dependence or abuse
* liver or kidney disease
* physician directed narcotic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 6 months
  VAS score for pain control, daily for two weeks post op and at all follow up visits for 6 months.
Narcotic Use | 2 months
  Measurement of both daily narcotic use in milligrams as well as the duration of narcotic treatment in days.
Patient Satisfaction | 3 months
  Measurement of patient satisfaction with pain control regimen using the American Pain Society's Patient Outcome Questionnaire (APS-POQ).

SECONDARY OUTCOMES:
Patient function | 6 months
  Measurement of patient function using the Short Musculoskeletal Functional Assessment questionnaire.
Fracture Union | 6 months
  Binary determination of fracture union (yes or no) during the 6 month duration of the study.
Adverse events | 6 months
  Measurement of the rate of adverse events post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Ostrum, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898
- [Background] Maheshwari AV, Boutary M, Yun AG, Sirianni LE, Dorr LD. Multimodal analgesia without routine parenteral narcotics for total hip arthroplasty. Clin Orthop Relat Res. 2006 Dec;453:231-8. doi: 10.1097/01.blo.0000246545.72445.c4. PMID 17031312
- [Background] Kashefi P, Honarmand A, Safavi M. Effects of preemptive analgesia with celecoxib or acetaminophen on postoperative pain relief following lower extremity orthopedic surgery. Adv Biomed Res. 2012;1:66. doi: 10.4103/2277-9175.100197. Epub 2012 Aug 28. PMID 23459777
- [Background] Panah Khahi M, Yaghooti AA, Marashi SH, Nadjafi A. Effect of pre-emptive gabapentin on postoperative pain following lower extremity orthopaedic surgery under spinal anaesthesia. Singapore Med J. 2011 Dec;52(12):879-82. PMID 22159930
- [Background] Montazeri K, Kashefi P, Honarmand A. Pre-emptive gabapentin significantly reduces postoperative pain and morphine demand following lower extremity orthopaedic surgery. Singapore Med J. 2007 Aug;48(8):748-51. PMID 17657384
- [Background] Ho KY, Gan TJ, Habib AS. Gabapentin and postoperative pain--a systematic review of randomized controlled trials. Pain. 2006 Dec 15;126(1-3):91-101. doi: 10.1016/j.pain.2006.06.018. Epub 2006 Jul 18. PMID 16846695
- [Background] Yadeau JT, Paroli L, Kahn RL, Jules-Elysee KM, Lasala VR, Liu SS, Lin E, Powell K, Buschiazzo VL, Wukovits B, Roberts MM, Levine DS. Addition of pregabalin to multimodal analgesic therapy following ankle surgery: a randomized double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2012 May-Jun;37(3):302-7. doi: 10.1097/AAP.0b013e31824c6846. PMID 22476240
- [Background] Khalili G, Janghorbani M, Saryazdi H, Emaminejad A. Effect of preemptive and preventive acetaminophen on postoperative pain score: a randomized, double-blind trial of patients undergoing lower extremity surgery. J Clin Anesth. 2013 May;25(3):188-92. doi: 10.1016/j.jclinane.2012.09.004. Epub 2013 Apr 6. PMID 23567482
- [Background] Rajpal S, Gordon DB, Pellino TA, Strayer AL, Brost D, Trost GR, Zdeblick TA, Resnick DK. Comparison of perioperative oral multimodal analgesia versus IV PCA for spine surgery. J Spinal Disord Tech. 2010 Apr;23(2):139-45. doi: 10.1097/BSD.0b013e3181cf07ee. PMID 20375829
- [Background] Hebl JR, Dilger JA, Byer DE, Kopp SL, Stevens SR, Pagnano MW, Hanssen AD, Horlocker TT. A pre-emptive multimodal pathway featuring peripheral nerve block improves perioperative outcomes after major orthopedic surgery. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):510-7. PMID 19258965
- [Background] Cho CH, Song KS, Min BW, Lee KJ, Ha E, Lee YC, Lee YK. Multimodal approach to postoperative pain control in patients undergoing rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2011 Oct;19(10):1744-8. doi: 10.1007/s00167-010-1294-y. Epub 2010 Oct 19. PMID 20957469
- [Background] Goldstein RY, Montero N, Jain SK, Egol KA, Tejwani NC. Efficacy of popliteal block in postoperative pain control after ankle fracture fixation: a prospective randomized study. J Orthop Trauma. 2012 Oct;26(10):557-61. doi: 10.1097/BOT.0b013e3182638b25. PMID 22732860
- [Background] VanDenKerkhof EG, Hopman WM, Goldstein DH, Wilson RA, Towheed TE, Lam M, Harrison MB, Reitsma ML, Johnston SL, Medd JD, Gilron I. Impact of perioperative pain intensity, pain qualities, and opioid use on chronic pain after surgery: a prospective cohort study. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):19-27. doi: 10.1097/AAP.0b013e318237516e. PMID 22157741
- [Background] Carroll I, Barelka P, Wang CK, Wang BM, Gillespie MJ, McCue R, Younger JW, Trafton J, Humphreys K, Goodman SB, Dirbas F, Whyte RI, Donington JS, Cannon WB, Mackey SC. A pilot cohort study of the determinants of longitudinal opioid use after surgery. Anesth Analg. 2012 Sep;115(3):694-702. doi: 10.1213/ANE.0b013e31825c049f. Epub 2012 Jun 22. PMID 22729963
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Remerand F, Le Tendre C, Baud A, Couvret C, Pourrat X, Favard L, Laffon M, Fusciardi J. The early and delayed analgesic effects of ketamine after total hip arthroplasty: a prospective, randomized, controlled, double-blind study. Anesth Analg. 2009 Dec;109(6):1963-71. doi: 10.1213/ANE.0b013e3181bdc8a0. PMID 19923527
- [Background] Ayalon O, Liu S, Flics S, Cahill J, Juliano K, Cornell CN. A multimodal clinical pathway can reduce length of stay after total knee arthroplasty. HSS J. 2011 Feb;7(1):9-15. doi: 10.1007/s11420-010-9164-1. Epub 2010 May 22. PMID 22294952
- [Background] Fu PL, Xiao J, Zhu YL, Wu HS, Li XH, Wu YL, Qian QR. Efficacy of a multimodal analgesia protocol in total knee arthroplasty: a randomized, controlled trial. J Int Med Res. 2010 Jul-Aug;38(4):1404-12. doi: 10.1177/147323001003800422. PMID 20926013
- [Background] Ho KY, Tay W, Yeo MC, Liu H, Yeo SJ, Chia SL, Lo NN. Duloxetine reduces morphine requirements after knee replacement surgery. Br J Anaesth. 2010 Sep;105(3):371-6. doi: 10.1093/bja/aeq158. Epub 2010 Jun 23. PMID 20573635
- [Background] Rasmussen ML, Mathiesen O, Dierking G, Christensen BV, Hilsted KL, Larsen TK, Dahl JB. Multimodal analgesia with gabapentin, ketamine and dexamethasone in combination with paracetamol and ketorolac after hip arthroplasty: a preliminary study. Eur J Anaesthesiol. 2010 Apr;27(4):324-30. doi: 10.1097/EJA.0b013e328331c71d. PMID 19734790
- [Background] Huang YM, Wang CM, Wang CT, Lin WP, Horng LC, Jiang CC. Perioperative celecoxib administration for pain management after total knee arthroplasty - a randomized, controlled study. BMC Musculoskelet Disord. 2008 Jun 3;9:77. doi: 10.1186/1471-2474-9-77. PMID 18519002
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Aida S, Fujihara H, Taga K, Fukuda S, Shimoji K. Involvement of presurgical pain in preemptive analgesia for orthopedic surgery: a randomized double blind study. Pain. 2000 Feb;84(2-3):169-73. doi: 10.1016/s0304-3959(99)00196-7. PMID 10666521
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Woodside JR. Female smokers have increased postoperative narcotic requirements. J Addict Dis. 2000;19(4):1-10. doi: 10.1300/J069v19n04_01. PMID 11110060
- [Background] Gorocs TS, Lambert M, Rinne T, Krekler M, Modell S. Efficacy and tolerability of ready-to-use intravenous paracetamol solution as monotherapy or as an adjunct analgesic therapy for postoperative pain in patients undergoing elective ambulatory surgery: open, prospective study. Int J Clin Pract. 2009 Jan;63(1):112-20. doi: 10.1111/j.1742-1241.2008.01914.x. PMID 19125998
- [Background] He BJ, Tong PJ, Li J, Jing HT, Yao XM. Auricular acupressure for analgesia in perioperative period of total knee arthroplasty. Pain Med. 2013 Oct;14(10):1608-13. doi: 10.1111/pme.12197. Epub 2013 Jul 18. PMID 23865512